CLINICAL TRIAL: NCT01385163
Title: Study of Intervention Effectiveness in Improving Psychosocial and Economic Well-being of Sexual Violence Survivors in DRC
Brief Title: Intervention Effectiveness in Improving Psychosocial and Economic Well-being of Sexual Violence Survivors in DRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JHU-AMHR-IRC-2010
Record Dates: First submitted 2011-06-22; First posted 2011-06-29 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Depression; Anxiety; PTSD
Keywords: mental health; gender-based violence; Africa
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 405+
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control - VSLA (No Intervention): the wait control sample for the economic intervention
- Control - Mental Health (Other): treatment as usual based on standard psychosocial services in the area
  Interventions: Behavioral: Treatment as usual
- Voluntary Savings/Loans Assoc (Experimental)
  Interventions: Behavioral: Voluntary Savings/Loans Assoc
- Cognitive Processing Therapy (Experimental)
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Treatment as usual — Standard psychosocial counseling
  Other Names: TAU
  Arms: Control - Mental Health
Behavioral: Voluntary Savings/Loans Assoc — economic intervention for group savings and loans
  Other Names: economic intervention of savings and loans program
  Arms: Voluntary Savings/Loans Assoc
Behavioral: Cognitive Processing Therapy — group 12 session intervention
  Other Names: cognitive behavioral therapy
  Arms: Cognitive Processing Therapy

SUMMARY:
The Democratic Republic of the Congo (DRC) has become synonymous with sexual violence by armed groups within the last 2 decades. Reportedly, tens of thousands of women and girls have been raped, sexually assaulted, attacked and abducted in the Eastern Provinces including North and South Kivu, targeted by armed groups with unparalleled levels of brutality.

Access to services in North and South Kivu-both emergency and longer term care-remains a major challenge. Limited services as well as the potential stigma of seeking services mean that many survivors have never received adequate care. Results of a preliminary study found many survivors have substantially reduced ability to function, including reduced ability to perform basic tasks and activities related to earning, self care, caring for family, and contributing to their communities. These survivors also describe high rates of mental health and social problems including mood disorders, anxiety, withdrawal, and stigmatization and rejection by family and community.

While social and economic development in conflict affected areas like DRC relies on populations who are ready and able to work, the psychological effects of conflict may mean that a percentage of the population living in these low-resource areas are less able to engage in economic opportunities even when they are available. However, there is little data on the best strategy to deal with this.

This study will be run as two parallel randomized impact evaluations to investigate the impacts of two different intervention programs to be implemented as part of standard programming of the collaborating NGO. The first study will focus on the impact of IRC's social-economic intervention, Village Savings and Loans Associations (VSLA) compared to a wait-control sample. The VSLA impact evaluation study will be conducted in communities served by 9 community-based organization (CBO) partners. The second study will focus on the impact of a mental health intervention, Cognitive Processing Therapy (CPT) compared to a wait-control sample. The CPT impact evaluation study will be conducted in communities serviced by NGO partners currently providing psychosocial support. As an exploratory investigation, the researchers will follow the CPT program with the VSLA program to look at the effect of receiving a mental health intervention prior to the VSLA on rates of retention and impact.

DETAILED DESCRIPTION:
These 2 parallel randomized controlled trials will use the same inclusion criteria and same assessments, but will have some differences in recruitment and program implementation periods.

For the mental health study, women will be recruited and then will initiate a 12-week treatment period when they will attend group sessions weekly with a trained counselor. Following the treatment period, a brief qualitative assessment will be conducted followed by a quantitative follow up of the intervention participants and wait-controls. A maintenance period of approximately 4 months will then begin when neither the intervention nor control participants will get any additional services from the counselors. Following the maintenance period, the intervention and control participants will again be assessed. If the intervention is found to be effective, the control counselors will be trained in the intervention and the controls will begin to receive the intervention. The original intervention participants, having successfully completed the mental health intervention, will then be invited to participate in the social-economic intervention. That program will begin within 1-2 months after the maintenance period is complete. The social-economic program (VSLA) will last approximately 9 months, after which the intervention participants will again be assessed.

For the VSLA study, eligible women will be recruited and invited to form groups to participate in the social-economic program (VSLA). Once eligibility is determined, the time to initiation of the VSLA program will be about 1 month. The VSLA program will include 8-10 weeks of active training with weekly or bi-weekly sessions, followed by a period of program implementation when the groups of women will save and make loans. At the end of 9 months, the women will complete the VSLA program cycle and get the financial returns on their funds. At that time, a brief qualitative assessment will be conducted followed by a quantitative assessment with the VSLA participants and controls. After the assessment, the control participants will be invited to participate in the VSLA program. All participants will then again be assessed when the controls have completed their program, after approximately 9 months.

ELIGIBILITY:
Inclusion Criteria:

* survivor of sexual violence
* mental health symptom severity cut-off
* functional impairment cut-off

Exclusion Criteria:

* active suicidality
* not living in the study site

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Severity of mental health symptoms | previous 4 weeks
  Several measures of mental health problems including depression, anxiety, and post-traumatic distress, will be assessed as primary outcomes.

SECONDARY OUTCOMES:
Economic development | prior 4 weeks
  A variety of economic indicators, including income, time spent working and food consumption, will be assessed for intervention impact.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Bass, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Village based, Bukavu, South Kivu, Democratic Republic of the Congo

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Murray SM, Augustinavicius J, Kaysen D, Rao D, Murray LK, Wachter K, Annan J, Falb K, Bolton P, Bass JK. The impact of Cognitive Processing Therapy on stigma among survivors of sexual violence in eastern Democratic Republic of Congo: results from a cluster randomized controlled trial. Confl Health. 2018 Feb 12;12:1. doi: 10.1186/s13031-018-0142-4. eCollection 2018. PMID 29449879
- [Derived] Bass JK, Annan J, McIvor Murray S, Kaysen D, Griffiths S, Cetinoglu T, Wachter K, Murray LK, Bolton PA. Controlled trial of psychotherapy for Congolese survivors of sexual violence. N Engl J Med. 2013 Jun 6;368(23):2182-91. doi: 10.1056/NEJMoa1211853. PMID 23738545